CLINICAL TRIAL: NCT01140477
Title: A Prospective Multicenter Clinical Trial To Evaluate the Effectiveness of A Toric Accommodating Posterior Chamber Silicone Intraocular Lens Designed To Provide Near, Intermediate, And Distance Vision And Reduce The Effects Of Preoperative Corneal Astigmatism On Postoperative Refraction Following Cataract Surgery
Brief Title: Toric Intraocular Lens Following Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 650
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism | interventions — Multifocal Intraocular Lenses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crystalens toric IOL (Experimental): Toric Accommodating Lens Crystalens toric silicone multi-piece accommodating IOL (Models AT-50T/AT-52T)
  Interventions: Device: Toric Accommodating Lens
- Crystalens IOL (Active Comparator): Accommodating Lens Crystalens silicone multi-piece accommodating IOL (Models AT-50SE/AT-52SE)
  Interventions: Device: Accommodating Lens

INTERVENTIONS:
Device: Toric Accommodating Lens — Toric accommodating lens implanted after cataract extraction
  Arms: Crystalens toric IOL
Device: Accommodating Lens — Accommodating lens implanted after cataract extraction
  Arms: Crystalens IOL

SUMMARY:
The objective of this clinical trial is to evaluate the safety and effectiveness of the Bausch + Lomb Toric Accommodating Posterior Chamber Silicone Intraocular Lens used to provide near, intermediate, and distance vision and a reduction of the effects of preoperative corneal astigmatism in presbyopic patients undergoing cataract extraction and intraocular lens (IOL) placement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented diagnosis of age-related cataract
* Subjects must require a lens power from 16 to 27 diopters
* Subjects must have predicted post-operative corneal astigmatism between 0.83D and 2.50D, as determined by the Toric Calculator

Exclusion Criteria:

* Subjects with any anterior segment pathology for which extracapsular/ phacoemulsification cataract surgery would be contraindicated.
* Subjects with diagnoses of degenerative visual disorders.
* Subjects with conditions associated with increased risk of zonular rupture.
* Subjects who have had previous corneal surgery in the planned operative eye.
* Subjects with irregular corneal astigmatism.
* Subjects with clinically significant retinal pigment or epithelium/macular changes.
* Subjects with chronic use of systemic steroids or immunosuppressive medications.
* Subjects either concurrently participating in another clinical trial or have participated in another clinical trial within 60 days prior to enrollment in this study.
* Subjects with a difference in corneal astigmatism measured with the IOL Master and the topographer greater than 0.5 D using vector analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pepose, MD, PhD, Study Director — Pepose Vision Institute
Locations (1):
- B&L Surgical, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crystalens Toric IOL: Crystalens toric silicone multi-piece accommodating IOL (Models AT-50T/AT-52T)
- Crystalens IOL: Crystalens silicone multi-piece accommodating IOL (Models AT-50SE/AT-52SE)
Period: Overall Study
Arm/Group | Crystalens Toric IOL | Crystalens IOL
Started | 153 | 76
Completed | 145 | 70
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Surgical complication preventing implant | 2 | 0
Not completed — Death | 1 | 1
Not completed — Subject explanted | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crystalens Toric IOL | Crystalens IOL | Total
Number analyzed (Participants) | 153 | 76 | 229
Age, Continuous [Mean (Full Range); unit: years] | 70.1 (9.0) [48 to 89] | 69.8 (9.2) [47 to 89] | 70.0 [47 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 42 | 123
  Male | 72 | 34 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Absolute Cylinder
Description: Percent reduction in absolute cylinder expressed as a percentage of the intended reduction in cylinder. Cylinder reduction is the measurement for astigmatism reduction. Astigmatism is a form of refractive error that can affect uncorrected visual acuity (at all distances). Reducing cylinder should improve UCVA, but other elements of refractive error, such as myopia or hyperopia, can also affect UCVA. Best corrected visual acuity (BCVA) is not affected by refractive error.
Time Frame: 120 - 180 day postoperative visit
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Mean (95% Confidence Interval); unit: percentage of intended cylinder reduct
Groups:
- Crystalens Toric IOL: Crystalens toric silicone multi-piece accommodating IOL (Models AT-50T/AT-52T)
  Toric Accommodating Lens: Toric accommodating lens implanted during cataract extraction
- Crystalens IOL: Crystalens silicone multi-piece accommodating IOL (Models AT-50SE/AT-52SE)
  Accommodating Lens: Accommodating lens implanted during cataract extraction
Arm/Group | Crystalens Toric IOL | Crystalens IOL
Number analyzed (Participants) | 134 | 68
percentage of intended cylinder reduct | 84.975 [79.961 to 89.989] | 46.498 [35.891 to 57.105]

2. Secondary Outcome: Lens Misalignment
Description: This Outcome Measure was evaluated for Crystalens Toric IOL arm only - Toric IOLs require precise alignment to correct astigmatism; control IOLs do not.
Time Frame: 120 - 180 day postoperative visit
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Crystalens Toric IOL
Number analyzed (Participants) | 130
degrees | 4.660 (4.208)

3. Secondary Outcome: Visual Acuity
Description: Best-Corrected Distance Visual Acuity (BCDVA) without Glare (logMAR)
Time Frame: 120 - 180 day postoperative visit
Population: The analysis population only includes those for whom the outcome was measured within the specified time frame.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Crystalens Toric IOL | Crystalens IOL
Number analyzed (Participants) | 134 | 68
logMAR | 0.004 (0.097) | 0.012 (0.094)

ADVERSE EVENTS:
Arm/Group | Crystalens Toric IOL | Crystalens IOL
Serious Adverse Events (participants affected / at risk) | 16/153 | 6/76
Other Adverse Events (participants affected / at risk) | 47/153 | 29/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalens Toric IOL (N=153) | Crystalens IOL (N=76)
Bronchopulmonary aspergillosis allergic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
High grade B-cell lymphoma, Burkitt-like lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bone sarcoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystalens Toric IOL (N=153) | Crystalens IOL (N=76)
Dry eye (Eye disorders) | 14 (26) | 3 (6)
Vitreous detachment (Eye disorders) | 17 (24) | 5 (8)
Blepharitis (Eye disorders) | 9 (17) | 4 (11)
Corneal oedema (Eye disorders) | 10 (16) | 2 (2)
Keratoconjunctivitis sicca (Eye disorders) | 6 (9) | 9 (15)
Conjunctivitis allergic (Eye disorders) | 3 (5) | 6 (10)
Punctate keratitis (Eye disorders) | 6 (9) | 4 (7)
Vitreous floaters (Eye disorders) | 6 (10) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of ten years, the PI agrees to keep confidential and not disclose, without the prior written consent of Sponsor, to any third party or use any technology, data, reports, results of clinical studies conducted under this Study or other information received by Sponsor, or any technology, data, reports, study materials, or other information developed by Sponsor unless disclosure by PI is required by law.